CLINICAL TRIAL: NCT00479713
Title: A Randomized, Double-Blind, Active-Controlled, Multicenter Study to Assess the LDL-C Lowering of Switching to a Combo Tab Ezetimibe/Simvastatin (10 mg/20 mg) Compared to Rosuvastatin 10 mg in Patients With Primary High Cholesterol and High Cardiovascular Risk Not Controlled With a Prior Statin Treatment
Brief Title: A Study to Assess the Cholesterol Lowering Effect of an Ezetimibe/Simvastatin Combination Tablet Compared to Another Cholesterol Lowering Drug in Patients With High Cholesterol and With High Cardiovascular Risk (0653A-809)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-809; 2007_552
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Results first posted 2009-06-10 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
Keywords: High Cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Arm 1: drug
  Interventions: Drug: ezetimibe (+) simvastatin; Drug: Comparator: Placebo (unspecified)
- 2 (Active Comparator): Arm 2: active comparator
  Interventions: Drug: Comparator : rosuvastatin calcium; Drug: Comparator: Placebo (unspecified)

INTERVENTIONS:
Drug: ezetimibe (+) simvastatin — ezetimibe/simvastatin 10/20mg. The treatment duration will be 6 weeks.
  Other Names: MK0653A; Vytorin®
  Arms: 1
Drug: Comparator : rosuvastatin calcium — rosuvastatin 10mg. The treatment duration will be 6 weeks.
  Arms: 2
Drug: Comparator: Placebo (unspecified) — rosuvastatin 10mg Placebo. The treatment duration will be 6 weeks.
  Arms: 1
Drug: Comparator: Placebo (unspecified) — ezetimibe/simvastatin 10/20mg Placebo. The treatment duration will be 6 weeks.
  Arms: 2

SUMMARY:
This is a multicenter study to evaluate the safety and efficacy of ezetimibe/simvastatin versus rosuvastatin in participants with high cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Participant is currently taking a statin medication for the treatment of high cholesterol
* Participant has an LDL-C level that is greater than or equal to 100 mg/dl and less than or equal to 190 mg/dl

Exclusion Criteria:

* Women who are pregnant or nursing, or women who intend to become pregnant
* Participant has any condition, situation, or is currently taking any medication that might pose a risk to the participant or interfere with participation in the study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 2007-02-01 (Actual); Primary Completion 2008-03-01 (Actual); Study Completion 2008-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farnier M, Averna M, Missault L, Vaverkova H, Viigimaa M, Massaad R, Vandormael K, Johnson-Levonas AO, Brudi P. Lipid-altering efficacy of ezetimibe/simvastatin 10/20 mg compared with rosuvastatin 10 mg in high-risk hypercholesterolaemic patients inadequately controlled with prior statin monotherapy - The IN-CROSS study. Int J Clin Pract. 2009 Apr;63(4):547-59. doi: 10.1111/j.1742-1241.2009.02022.x. Epub 2009 Feb 16. PMID 19222610
- [Derived] Averna M, Missault L, Vaverkova H, Farnier M, Viigimaa M, Dong Q, Shah A, Johnson-Levonas AO, Taggart W, Brudi P. Lipid-altering efficacy of switching to ezetimibe/simvastatin 10/20 mg versus rosuvastatin 10 mg in high-risk patients with and without metabolic syndrome. Diab Vasc Dis Res. 2011 Oct;8(4):262-70. doi: 10.1177/1479164111418136. Epub 2011 Aug 22. PMID 21859750
- [Derived] Viigimaa M, Vaverkova H, Farnier M, Averna M, Missault L, Hanson ME, Dong Q, Shah A, Brudi P. Ezetimibe/simvastatin 10/20 mg versus rosuvastatin 10 mg in high-risk hypercholesterolemic patients stratified by prior statin treatment potency. Lipids Health Dis. 2010 Nov 4;9:127. doi: 10.1186/1476-511X-9-127. PMID 21050476

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase IV
  First Participant In: 31-Mar-2007; Last Participant Last Visit 11-Mar-2008
  85 centers worldwide (EX US)
  Eligible participants include those on a stable dose of one of the following: rosuvastatin 5 mg; simvastatin 20 mg, 40 mg; atorvastatin 10, 20 mg; pravastatin 40 mg; fluvastatin 80 mg.
Pre-assignment Details: Eligible participants were randomized at Visit 2 (Week 6) to either a combination tablet of ezetimibe/simvastatin (10 mg/20 mg) plus a matching placebo for rosuvastatin 10 mg (Group 1) or rosuvastatin 10 mg plus a matching placebo for the combination tablet (Group 2) for a 6-week treatment period.
Groups:
- Ezetemibe + Simvastatin: Ezetemibe 10 mg + Simvastatin 20 mg plus a matching placebo for rosuvastatin 10 mg QD (once a day) for 6 weeks
- Rosuvastatin: Rosuvastatin 10 mg plus a matching placebo for the combination tablet QD (once a day) for 6 weeks
Period: Overall Study
Arm/Group | Ezetemibe + Simvastatin | Rosuvastatin
Started | 314 | 304
Completed | 301 | 295
Not Completed | 13 | 9
Not completed — Adverse Event | 8 | 6
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetemibe + Simvastatin | Rosuvastatin | Total
Number analyzed (Participants) | 314 | 304 | 618
Age, Continuous [Mean (Full Range); unit: years] | 63.2 [38 to 82] | 63.1 [27 to 80] | 63.15 [27 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 119 | 248
  Male | 185 | 185 | 370
Race/Ethnicity, Customized [Number; unit: participants]
  White | 314 | 302 | 616
  Black | 0 | 2 | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 37 | 43 | 80
  Not Hispanic or Latino | 277 | 261 | 538
Apolipoprotein B [Median (Standard Deviation); unit: mg/dL] | 1.20 (0.20) | 1.18 (0.21) | 1.19 (0.21)
C Reactive Protein [Median (Standard Deviation); unit: mg/dL] | 0.16 (0.26) | 0.15 (0.26) | 0.16 (0.26)
High Density Lipoprotein-Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 1.43 (0.37) | 1.43 (0.36) | 1.43 (0.36)
Low Density Lipoprotein-Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 3.21 (0.42) | 3.24 (0.44) | 3.23 (0.43)
Low Density Lipoprotein-Cholesterol (LDL-C):High Density Lipoprotein-Cholesterol (HDL-C) ratio [Mean (Standard Deviation); unit: LDL-C:HDL-C ratio] | 2.38 (0.65) | 2.40 (0.65) | 2.39 (0.65)
Non-High Density Lipoprotein-Cholesterol (Non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 3.95 (0.55) | 3.95 (0.56) | 3.95 (0.55)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 5.38 (0.57) | 5.38 (0.61) | 5.38 (0.59)
Total cholesterol:High Density Lipoprotein-Cholesterol (HDL-C) ratio [Mean (Standard Deviation); unit: Total cholesterol:HDL-C ratio] | 3.94 (0.89) | 3.96 (0.90) | 3.95 (0.90)
Triglycerides [Median (Standard Deviation); unit: mg/dL] | 1.46 (0.86) | 1.41 (0.87) | 1.42 (0.88)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Low Density Lipoprotein-Cholesterol (LDL-C) at Study Endpoint After Six Weeks of Treatment
Description: Percent Change in LDL-C at study endpoint after six weeks of treatment is calculated as the difference between week 6 measure and baseline measure divided by baseline measure *100.
Time Frame: Baseline and 6 weeks
Population: Full Analysis Set (FAS): The FAS population includes all randomized participants who took at least 1 dose of study medication and had a baseline (BL) value and at least one post BL value.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetemibe + Simvastatin | Rosuvastatin
Number analyzed (Participants) | 305 | 297
percent change from baseline | -27.66 [-30.27 to -25.04] | -16.94 [-19.61 to -14.28]
Statistical Analysis 1: Comparison: Ezetemibe + Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p <= 0.001, ANOVA; Model terms: treatment, stratum, baseline (categorized based on quartiles) and center; Mean Difference (Final Values) = -10.72, 95% CI [-14.10 to -7.33], Standard Error of Mean 1.72

2. Secondary Outcome: The Percentage of Participants Achieving Designated Low Density Lipoprotein-Cholesterol (LDL-C) Levels After 6 Weeks of Treatment
Description: The percentage of participants who achieved a target LDL-C goal of < 100 mg/dL, of <70 mg/dL, and of <77 mg/dL at study endpoint after six weeks of treatment.
  The numerator is the number of participants in a treatment group who achieved a target LDL-C goal and the denominator is the total number of participants within that treatment group.
Time Frame: after 6 weeks of treatment
Population: Full Analysis Set (FAS)
Measure: Number; unit: Percent of participant population
Arm/Group | Ezetemibe + Simvastatin | Rosuvastatin
Number analyzed (Participants) | 305 | 297
Percent of participant population
  LDL-C <100 | 72.46 | 56.23
  LDL-C <70 | 25.25 | 11.11
Statistical Analysis 1: Comparison: Ezetemibe + Simvastatin vs Rosuvastatin; Percentage of Participants who Attained Target LDL-C Goal of < 100 mg/dL (2.59 mmol/L); Test type: Superiority or Other; p <= 0.001, Regression, Logistic; Model terms: treatment, stratum and baseline LDL-C (continuous); Odds Ratio (OR) = 2.1, 95% CI [1.5 to 3.0]
Statistical Analysis 2: Comparison: Ezetemibe + Simvastatin vs Rosuvastatin; Percentage of Participants who Attained Target LDL-C Goal of < 70 mg/dL (1.81 mmol/L); Test type: Superiority or Other; p <= 0.001, Regression, Logistic; Model terms: treatment, stratum and baseline LDL-C (continuous); Odds Ratio (OR) = 2.8, 95% CI [1.8 to 4.4]

3. Other Pre Specified Outcome: Percent Change From Baseline in Total Cholesterol
Description: Percent change from baseline in total cholesterol at study endpoint after 6 weeks of treatment is calculated as the difference between week 6 measure and baseline measure divided by baseline measure *100.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetemibe + Simvastatin | Rosuvastatin
Number analyzed (Participants) | 305 | 297
percent change from baseline | -17.53 [-19.36 to -15.71] | -10.33 [-12.19 to -8.47]
Statistical Analysis 1: Comparison: Ezetemibe + Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p <= 0.001, ANOVA; Model terms: treatment, stratum, baseline (categorized based on quartiles) and center; Mean Difference (Final Values) = -7.20, 95% CI [-9.56 to -4.84], Standard Error of Mean 1.20

4. Other Pre Specified Outcome: Percent Change From Baseline in Triglycerides.
Description: Percent change from baseline in triglycerides at study endpoint after 6 weeks of treatment is calculated as the difference between week 6 measure and baseline measure divided by baseline measure *100.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetemibe + Simvastatin | Rosuvastatin
Number analyzed (Participants) | 305 | 297
percent change from baseline | -11.00 [-15.25 to -6.80] | -5.26 [-9.92 to -1.17]
Statistical Analysis 1: Comparison: Ezetemibe + Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.056, Nonparametric ANOVA; ANOVA model based on Tukey's normalized ranks with term for treatment, stratum, baseline (categorized based on quartiles) and center; Median Difference (Final Values) = -5.06, 95% CI [-9.56 to -0.30] — The median difference between treatments is based on the Hodges-Lehmann estimates of shift with a corresponding distribution-free Confidence Interval (CI) based on Wilcoxon's rank

5. Other Pre Specified Outcome: Percent Change From Baseline in High Density Lipoprotein-Cholesterol (HDL-C)
Description: Percent change from baseline in HDL-C at study endpoint after 6 weeks of treatment is calculated as the difference between week 6 measure and baseline measure divided by baseline measure *100.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetemibe + Simvastatin | Rosuvastatin
Number analyzed (Participants) | 305 | 297
percent change from baseline | 2.12 [0.34 to 3.89] | 3.03 [1.22 to 4.85]
Statistical Analysis 1: Comparison: Ezetemibe + Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.433, ANOVA; Model terms: treatment, stratum, baseline (categorized based on quartiles) and center; Mean Difference (Final Values) = -0.92, 95% CI [-3.21 to 1.38], Standard Error of Mean 1.17

6. Other Pre Specified Outcome: Percent Change From Baseline in Non-High Density Lipoprotein-Cholesterol (Non-HDL-C)
Description: Percent change from baseline in non HDL-C at study endpoint after 6 weeks of treatment is calculated as the difference between week 6 measure and baseline measure divided by baseline measure *100.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetemibe + Simvastatin | Rosuvastatin
Number analyzed (Participants) | 305 | 297
percent change from baseline | -23.42 [-25.81 to 21.03] | -14.01 [-16.46 to -11.57]
Statistical Analysis 1: Comparison: Ezetemibe + Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p <= 0.001, ANOVA; Model terms: treatment, stratum, baseline (categorized based on quartiles) and center; Mean Difference (Final Values) = -9.41, 95% CI [-12.50 to -6.31], Standard Error of Mean 1.58

7. Other Pre Specified Outcome: Percent Change From Baseline in Low Density Lipoprotein-Cholesterol (LDL-C)/High Density Lipoprotein-Cholesterol (HDL-C) Ratio
Description: Percent change from baseline in LDL-C/HDL-C ratio at study endpoint after 6 weeks of treatment is calculated as the difference between week 6 measure and baseline measure divided by baseline measure *100.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetemibe + Simvastatin | Rosuvastatin
Number analyzed (Participants) | 305 | 297
percent change from baseline | -27.41 [-30.42 to -24.40] | -17.82 [-20.89 to -14.75]
Statistical Analysis 1: Comparison: Ezetemibe + Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p <= 0.001, ANOVA; Model terms: treatment, stratum, baseline (categorized based on quartiles) and center; Mean Difference (Final Values) = -9.59, 95% CI [-13.49 to -5.69], Standard Error of Mean 1.98

8. Other Pre Specified Outcome: Percent Change From Baseline in Total Cholesterol/High Density Lipoprotein-Cholesterol (HDL-C) Ratio
Description: Percent change from baseline in total cholesterol/HDL-C ratio at study endpoint after 6 weeks of treatment is calculated as the difference between week 6 measure and baseline measure divided by baseline measure *100.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetemibe + Simvastatin | Rosuvastatin
Number analyzed (Participants) | 305 | 297
percent change from baseline | -17.76 [-19.94 to -15.57] | -11.51 [-13.74 to -9.28]
Statistical Analysis 1: Comparison: Ezetemibe + Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p <= 0.001, ANOVA; Model terms: treatment, stratum, baseline (categorized based on quartiles) and center; Mean Difference (Final Values) = -6.25, 95% CI [-9.07 to -3.43], Standard Error of Mean 1.44

9. Other Pre Specified Outcome: Percent Change From Baseline in Apolipoprotein B
Description: Percent change from baseline in apolipoprotein (Apo) B at study endpoint after 6 weeks of treatment is calculated as the difference between week 6 measure and baseline measure divided by baseline measure *100.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetemibe + Simvastatin | Rosuvastatin
Number analyzed (Participants) | 301 | 292
percent change from baseline | -17.87 [-20.05 to -15.70] | -9.77 [-11.99 to -7.55]
Statistical Analysis 1: Comparison: Ezetemibe + Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p <= 0.001, ANOVA; Model terms: treatment, stratum, baseline (categorized based on quartiles) and center; Mean Difference (Final Values) = -8.11, 95% CI [-10.91 to -5.30], Standard Error of Mean 1.43

10. Other Pre Specified Outcome: Percent Change From Baseline in High-sensitivity C (Hs-C) Reactive Protein
Description: Percent change from baseline in hs-C reactive protein at study endpoint after 6 weeks of treatment is calculated as the difference between week 6 measure and baseline measure divided by baseline measure *100.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Ezetemibe + Simvastatin | Rosuvastatin
Number analyzed (Participants) | 301 | 293
percent change from baseline | -8.33 [-16.67 to 0.00] | 0.00 [-7.14 to 6.25]
Statistical Analysis 1: Comparison: Ezetemibe + Simvastatin vs Rosuvastatin; Test type: Superiority or Other; p = 0.172, Nonparametric ANOVA; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -6.67, 95% CI [-16.67 to 2.87] — The median difference between treatments is based on the Hodges-Lehmann estimates of shift with a corresponding distribution-free CI based on Wilcoxon's rank

ADVERSE EVENTS:
Description: Adverse event tables include all participants who took at least one dose of study drug.
Arm/Group | Ezetemibe + Simvastatin | Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 3 | 5
Other Adverse Events (participants affected / at risk) | 19 | 30
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Ezetemibe + Simvastatin | Rosuvastatin
Cholangitis (Hepatobiliary disorders) | 1/312 | 0/304
Accidental overdose (Injury, poisoning and procedural complications) | 1/312 | 0/304
Subarachnoid hemorrhage (Nervous system disorders) | 1/312 | 0/304
Chest pain (General disorders) | 0/312 | 2/304
Epileptic seizure (Nervous system disorders) | 0/312 | 1/304
Skin eruption (Skin and subcutaneous tissue disorders) | 0/312 | 1/304
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 0/312 | 1/304
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Ezetemibe + Simvastatin | Rosuvastatin
Angina unstable (Cardiac disorders) | 1/312 | 0/304
Bradycardia (Cardiac disorders) | 1/312 | 0/304
Abdominal pain (Gastrointestinal disorders) | 2/312 | 2/304
Abdominal pain upper (Gastrointestinal disorders) | 1/312 | 1/304
Diarrhoea (Gastrointestinal disorders) | 3/312 | 1/304
Dry mouth (Gastrointestinal disorders) | 0/312 | 1/304
Dyspepsia (Gastrointestinal disorders) | 3/312 | 1/304
Nausea (Gastrointestinal disorders) | 2/312 | 0/304
Salivary hypersecretion (Gastrointestinal disorders) | 1/312 | 0/304
Vomitting (Gastrointestinal disorders) | 2/312 | 0/304
Asthenia (General disorders) | 0/312 | 1/304
Chest pain (General disorders) | 1/312 | 0/304
Pain (General disorders) | 0/312 | 1/304
Hypersensitivity (Immune system disorders) | 1/312 | 0/304
Seasonal allergy (Immune system disorders) | 1/312 | 0/304
Ear infection (Infections and infestations) | 0/312 | 1/304
Gastroenteritis (Infections and infestations) | 0/312 | 1/304
Gastroenteritis viral (Infections and infestations) | 0/312 | 1/304
Localised infection (Infections and infestations) | 0/312 | 1/304
Nasopharyngitis (Infections and infestations) | 1/312 | 0/304
Paronychia (Infections and infestations) | 0/312 | 1/304
Pharyngitis (Infections and infestations) | 1/312 | 0/304
Sinusitis (Infections and infestations) | 1/312 | 0/304
Tooth abscess (Infections and infestations) | 0/312 | 1/304
Contusion (Injury, poisoning and procedural complications) | 0/312 | 1/304
Deafness traumatic (Injury, poisoning and procedural complications) | 1/312 | 0/304
Fall (Injury, poisoning and procedural complications) | 1/312 | 0/304
Rib fracture (Injury, poisoning and procedural complications) | 1/312 | 0/304
Upper limb fracture (Injury, poisoning and procedural complications) | 0/312 | 1/304
Blood pressure increased (Investigations) | 0/312 | 1/304
Anorexia (Metabolism and nutrition disorders) | 1/312 | 0/304
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/312 | 1/304
Bursitis (Musculoskeletal and connective tissue disorders) | 0/312 | 1/304
Flank pain (Musculoskeletal and connective tissue disorders) | 1/312 | 0/304
Myalgia (Musculoskeletal and connective tissue disorders) | 3/312 | 2/304
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/312 | 0/304
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0/312 | 1/304
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/312 | 1/304
Carpal tunnel syndrome (Nervous system disorders) | 0/312 | 1/304
Headache (Nervous system disorders) | 1/312 | 0/304
Memory impairment (Nervous system disorders) | 0/312 | 1/304
Paraesthesia (Nervous system disorders) | 0/312 | 1/304
Syncope vasovagal (Nervous system disorders) | 0/312 | 1/304
Insomnia (Psychiatric disorders) | 0/312 | 1/304
Nervousness (Psychiatric disorders) | 0/312 | 1/304
Nephrolithiasis (Renal and urinary disorders) | 0/312 | 1/304
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0/312 | 1/304
Rash (Skin and subcutaneous tissue disorders) | 0/312 | 1/304
Hypertension (Vascular disorders) | 0/312 | 1/304
Bronchitis (Infections and infestations) | 2/312 | 0/304

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.